CLINICAL TRIAL: NCT04895514
Title: Use of Gamma-Irradiated Preserved Corneal Tissue to Treat Keratoconus
Brief Title: Gamma-Irradiated Corneal Inlay for Keratoconus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cornea and Laser Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAMMA TISSUE INLAY
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corneal tissue inlay (Experimental): The treated cornea will be implanted with a thin disc of gamma-irradiated preserved corneal tissue
  Interventions: Procedure: Gamma-irradiated corneal tissue inlay

INTERVENTIONS:
Procedure: Gamma-irradiated corneal tissue inlay — A mid-stomal pocket will be made into the cornea with a femtosecond laser (Intralase). A small disc of gamma-irradiated preserved corneal tissue will then be placed into the pocket

SUMMARY:
Study objective is to evaluate the outcomes of placing gamma-irradiated corneal tissue (VisionGraft, CorneaGen, USA) within the cornea of patients with keratoconus, a procedure called Corneal Tissue Addition for Keratoconus (CTAK).

DETAILED DESCRIPTION:
Using E gamma irradiated sterilized preserved corneal tissue, shaped corneal tissue inlays are placed in a keratoconic cornea. Preserved corneal tissue is currently available commercially from CorneaGen (VisionGraft,1200 6th Ave., STe.300, Seattle, WA 98101). Such tissue is currently used in a number of eye surgical procedures. It is considered suitable for corneal surgical procedures that do not require viable corneal endothelium, as is the case for a tissue enhancement procedure in keratoconus. The goal of the current protocol to evaluate the outcomes of placing gamma-irradiated preserved tissue within the keratoconic cornea in order to enhance corneal thickness, stability, and optical conformation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, male or female, of any race
* Provide written consent and sign a HIPAA form
* Willingness and ability to follow all instructions and comply with schedule for follow-up visits
* For females: must not be pregnant
* Having topographic evidence of keratoconus which is graded as moderate or severe keratoconus defined as the following:

  * Moderate Keratoconus: Axial topography consistent with keratoconus, Maximum keratometry on Pentacam greater than or equal to 51.01 D
  * Severe Keratoconus: Axial topography consistent with keratoconus with marked areas of steepening, Maximum keratometry on Pentacam greater than or equal to 56.01 D
* Presence of central or inferior steepening on the Pentacam map
* BSCVA less than or equal to 20/25
* Contact lens wearers only: remove contact lenses one week prior to the screening refraction

Exclusion Criteria:

* Contraindications, sensitivity or known allergy to the use of the test article(s) or their components
* If female, be pregnant
* Eyes classified as either normal, atypical normal, keratoconus suspect or mild keratoconus on the severity grading scheme
* Previous ocular condition (other than refractive error) in the eye to be treated that may predispose the eye for future complications. For example:

  a) History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, corneal melt, corneal dystrophy, etc.)
* A history of delayed epithelial healing in the eye to be treated
* Have used an investigational drug or device within 30 days of the study or be concurrently enrolled in another investigational drug or device study within 30 days of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Gamma-Irradiated Preserved Corneal Tissue Inlay | 6 months
  Change in mean keratometry on corneal topography

SECONDARY OUTCOMES:
Gamma Irradiated Preserved Corneal Tissue Inlay | 6 months
  Inferior-Superior (I-S) ratio
Gamma Irradiated Preserved Corneal Tissue Inlay | 6 months
  Manifest refraction
Gamma Irradiated Preserved Corneal Tissue Inlay | 6 months
  Uncorrected distance visual acuity
Gamma Irradiated Preserved Corneal Tissue Inlay | 6 months
  Best spectacle corrected distance visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Hersh, MD, Principal Investigator — Cornea and Laser Eye Institute; Steven A Greenstein, MD, Principal Investigator — Cornea and Laser Eye Institute
Locations (1):
- Cornea and Laser Eye Institute, Hersh Vision Group, Teaneck, New Jersey, United States